CLINICAL TRIAL: NCT04662918
Title: Validation of CAGIB Score for In-hospital Mortality of Cirrhotic Patients With Acute Gastrointestinal Bleeding: A Prospective, International Multicenter, Observational Study
Brief Title: Validation of CAGIB Score for In-hospital Mortality of Cirrhotic Patients With Acute Gastrointestinal Bleeding
Status: Recruiting | Type: Observational
Sponsor: Xingshun Qi (Other)
Responsible Party: Sponsor-Investigator, Xingshun Qi, Dr., Associate Professor, Vice-Chief Physician, General Hospital of Shenyang Military Region
Organization: General Hospital of Shenyang Military Region (Other)
Other Study IDs: V-CAGIB 1.0
Record Dates: First submitted 2020-12-02; First posted 2020-12-10 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: GastroIntestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Acute gastrointestinal bleeding is potentially lethal in liver cirrhosis. Accurate assessment of prognosis is critical in a timely fashion. A novel model, CAGIB score, has been developed based on our Chinese multicenter retrospective study. Now, a prospective, international multicenter, observational study will be performed to further compare the performance of CAGIB versus Child-Pugh and MELD scores for evaluating the in-hospital mortality of patients with liver cirrhosis and acute gastrointestinal bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with liver cirrhosis;
2. Patients with acute gastrointestinal bleeding presenting with hematemesis, melena, and/or hematochezia;
3. Adults (age≥18 years old).

Exclusion Criteria:

1. Components of Child-Pugh, MELD, and CAGIB scores are not available;
2. In-hospital outcomes are not evaluable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis and acute gastrointestinal bleeding
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | An average of 1-6 weeks, from admission to discharge
  Death caused by any events during hospitalizations.

SECONDARY OUTCOMES:
Failure to control bleeding within 5 days | 5 days
  Failure is defined as death or need to change therapy defined by one of the following criteria within 5 days: 1) Fresh hematemesis or nasogastric aspiration of ≥100 ml of fresh blood ≥2 h after the start of a specific drug treatment or therapeutic endoscopy; 2) Development of hypovolaemic shock; 3) 3g drop in hemoglobin (9% drop of hematocrit) within any 24 hours period if no transfusion is administered.

CONTACTS AND LOCATIONS:
Locations (23):
- The Wright Center for Graduate Medical Education, 501 S. Washington Avenue, Scranton, Pennsylvania, United States
- São Paulo State University (UNESP), Botucatu Medical School, São Paulo, São Paulo, Brazil
- China (16):
  - Beijing Youan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Seventh Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Six People's Hospital of Dalian, Dalian, Liaoning
  - Air Force Hospital of Northern Theater Command, Shenyang, Liaoning
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Six People's Hospital of Shenyang, Shenyang, Liaoning
  - Tangdu Hospital, Fourth Military Medical University,, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi
  - The Second Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi
  - Xi'an Central Hospital, Xi'an, Shaanxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - Cathay General Hospital, Fu-Jen Catholic University School of Medicine, Taibei, Taiwan
- Charité University Medical Center, Berlin, State of Berlin, Germany
- Ernakulam Medical Center, Kochi, Kochi, India
- Azienda di Rilievo Nazionale ad Alta Specializzazione Civico-Di Cristina-Benfratelli, Palermo, Palermo, Italy
- National Autonomous University of Mexico, Mexico City, Mexico City, Mexico
- Bezmialem Vakif University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bai Z, Li B, Lin S, Liu B, Li Y, Zhu Q, Wu Y, Yang Y, Tang S, Meng F, Chen Y, Yuan S, Shao L, Qi X. Development and Validation of CAGIB Score for Evaluating the Prognosis of Cirrhosis with Acute Gastrointestinal Bleeding: A Retrospective Multicenter Study. Adv Ther. 2019 Nov;36(11):3211-3220. doi: 10.1007/s12325-019-01083-5. Epub 2019 Sep 11. PMID 31512140
- [Derived] Zhang S, Sun M, Yuan S, Lin S, Romeiro FG, He Y, Zhu Q, Ma D, Li Y, Philips CA, Liu X, Mendez-Sanchez N, Shao L, Wu Y, Basaranoglu M, Pinyopornpanish K, Chen Y, Mancuso A, Yang L, Tacke F, Li B, Liu L, Ji F, Qi X. Identifying Low-Risk Patients with Cirrhosis and Acute Gastrointestinal Bleeding That May Not Require Urgent Endoscopy. Adv Ther. 2025 Nov 22. doi: 10.1007/s12325-025-03395-1. Online ahead of print. PMID 41273618
- [Derived] Bai Z, Lin S, Sun M, Yuan S, Marcondes MB, Ma D, Zhu Q, Li Y, He Y, Philips CA, Liu X, Pinyopornpanish K, Shao L, Mendez-Sanchez N, Basaranoglu M, Wu Y, Chen Y, Yang L, Mancuso A, Tacke F, Li B, Liu L, Ji F, Qi X. Machine learning based CAGIB score predicts in-hospital mortality of cirrhotic patients with acute gastrointestinal bleeding. NPJ Digit Med. 2025 Jul 31;8(1):489. doi: 10.1038/s41746-025-01883-w. PMID 40745090
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31512140/